CLINICAL TRIAL: NCT00594308
Title: In-Vivo Activated T-Cell Depletion to Prevent GVHD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Treatment ineffective
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0705-20 IUCRO-0196
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Results first posted 2012-03-20 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-09

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphocytic Leukemia; Chronic Myelogenous Leukemia; Chronic Lymphocytic Leukemia; Myelodysplasia; Lymphoma, Non-Hodgkin's; Mantle-Cell Lymphoma; Hodgkin's Disease; Multiple Myeloma; Myelofibrosis
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Anemia, Refractory, with Excess of Blasts; Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell; Hodgkin Disease; Multiple Myeloma; Primary Myelofibrosis | interventions — Cyclophosphamide; fludarabine; Cyclosporine; Mycophenolic Acid; Basiliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cyclophosphamide — 60mg/kg/day for two consecutive days (-7,-6).
Drug: Fludarabine — 25mg/m2/day for 5 consecutive days
Drug: Cyclosporine — 3mg/kg/day will be given by continuous intravenous infusion beginning on Day -1.
Drug: Mycophenolate mofetil — 1000 mg will be administered through day +60 and then discontinued if there is no GVHD.
Drug: Basiliximab — 20mg , will be given by intravenous infusion (without an in-line filter) over at least 15 minutes beginning 3 days after engraftment.

SUMMARY:
The purpose of this study is to compare the effects (good and bad) of the medication basiliximab in combination with cyclosporine with cyclosporine alone for the prevention of graft-versus-host disease.

This research is being done because there is no completely safe and effective prevention for graft-versus-host disease. It is known that cyclosporine helps with GVHD but we would like to know if the addition of basiliximab will decrease the incidence and/or severity of GVHD after a transplant known as nonmyeloablative ("mini" transplant).

ELIGIBILITY:
Inclusion Criteria:

* Acute myelogenous leukemia, Acute lymphocytic leukemia, Chronic myelogenous leukemia, Chronic lymphocytic leukemia, Myelodysplasia, Non-Hodgkin's Lymphoma, Mantle cell, Hodgkin's Disease, Multiple Myeloma, Myelofibrosis with disease-specific eligibility requirements as outlined in the protocol
* Donor Requirement: Must have a fully HLA-matched (10 of 10) related or unrelated donor, eighteen years of age or older, who is capable of undergoing GCSF mobilization and apheresis.

Exclusion Criteria:

* Active CNS disease (the presence of leukemic blasts in the CSF)
* Pregnancy or breast-feeding
* SGOT >3x upper limit of normal
* Creatinine >2 or creatinine clearance <50cc/hr.
* Fractional shortening by echocardiogram not within normal limits per institution
* Pulmonary function: DLCO less that 50% of normal predicted, corrected for anemia
* Prior allogeneic transplant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Nelson, MD, Principal Investigator — Indiana Universtiy School of Medicine
Locations (1):
- Indiana Universtiy Simon Cancer Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Basiliximab 20 mg: All patients that received Basiliximab 20 mg monoclonal therapy
Period: Overall Study
Arm/Group | Basiliximab 20 mg
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Basiliximab 20 mg
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.80 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Acute Grade II-IV GVHD
Description: Number of patients with Grade II-IV GVHD according to NMDP/CIBMTR GVHD severity scale. This scale measures the degree of GVHD involvement in the patient's skin (inflammatory skin disease), liver (bilirubin levels) and intestinal tract (amount of diarrhea) as well as the level of decline in a patient's activity and physical abilities.
Time Frame: until 30 days after stem cell transplant
Population: All patient that received study drug
Measure: Number; unit: participants
Arm/Group | Basiliximab 20 mg
Number analyzed (Participants) | 10
participants | 10

2. Secondary Outcome: Number of Patients Engrafting at Day +30 by Short Tandem Repeat (STR) on Peripheral Blood Mononuclear Cells (PBMC's).
Time Frame: until 30 days after stem cell transplant
Population: ITT population. All patient that received study drug
Measure: Number; unit: participants
Arm/Group | Basiliximab 20 mg
Number analyzed (Participants) | 10
participants | 10

3. Secondary Outcome: Number of Days for Absolute Neutrophil Count to Recover
Description: Average number of day per patient for absolute neutrophil count to recover(> 500/mm3 for 3 consecutive days).
Time Frame: From Day -1 (day before stem cell infusion) to Day+20 (20 days after stem cell infusion)
Population: ITT: All patient that received study drug
Measure: Mean (Standard Deviation); unit: days per patient
Arm/Group | Basiliximab 20 mg
Number analyzed (Participants) | 10
days per patient | 14.00 (3.80)

4. Secondary Outcome: Time to Resolution of Cytopenias: Platelet Transfusion Independence
Description: Average number of days per patient for resolution of cytopenias.
Time Frame: From Day -1 (day before stem cell infusion) to Day +20 (20 days after stem cell infusion)
Population: IIT: All patients that received study drug.
Measure: Mean (Standard Deviation); unit: days per patient
Arm/Group | Basiliximab 20 mg
Number analyzed (Participants) | 10
days per patient | 15.33 (3.54)

5. Secondary Outcome: Patients Who Experience Serious Transplant Related Toxicities as Evaluated by Bone Marrow Transplant-adjusted NCI Common Toxicity Criteria.
Description: Number of patients who died due to transplant related toxicities
Time Frame: up to 2 years after stem cell transplant
Population: Intent To Treat: All patients that received study drug
Measure: Number; unit: participants
Arm/Group | Basiliximab 20 mg
Number analyzed (Participants) | 10
participants | 10

ADVERSE EVENTS:
Arm/Group | Basiliximab 20 mg
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Basiliximab 20 mg (N=10)
GvHD (Immune system disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
Four patients experienced grade 3-4 GVHD and this study was stopped.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No